CLINICAL TRIAL: NCT02568709
Title: Effects of Oxytocin on Neural Activation Patterns During Social Cognitive Tasks in Patients With Schizophrenia
Brief Title: Oxytocin MEG Study
Acronym: MEG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12-08411
Record Dates: First submitted 2015-09-29; First posted 2015-10-06 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia; Oxytocin; Magnetoencephalography (MEG); Social Cognition
Keywords: Oxytocin; Syntocinon; Social Cognition; Schizophrenia; Magnetoencephalography (MEG)
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (Active Comparator): 40 IU Oxytocin
  Interventions: Drug: Oxytocin
- Saline Nasal Spray (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Saline Nasal Spray

INTERVENTIONS:
Drug: Oxytocin — 40 IU of the oxytocin will be administered intranasally for a one time dose at the beginning of the visit.
  Other Names: Syntocinon
  Arms: Interventional
Drug: Saline Nasal Spray — 40 IU of the saline nasal spray will be administered once at the beginning of the visit.
  Other Names: Placebo
  Arms: Saline Nasal Spray

SUMMARY:
The specific aim of this proposal is to investigate the neurophysiological mechanisms of oxytocin's (OT) prosocial effects in patients with schizophrenia and healthy subjects using magnetoencephalography.

Hypothesis A: When OT is administered to patients with schizophrenia, fear-related amygdala hyperreactivity and fusiform gyrus (FG) and anterior cingulate cortex (ACC) hypoactivity will be normalized.

Hypothesis B: When OT is administered to patients with schizophrenia, the decreased functional connectivity (FC) between the amygdala, FG, and ACC will be normalized.

By elucidating the neurophysiological mechanisms of OT administration on emotional face processing, investigators will bee able to:

1. understand the pathophysiology of the functionally debilitating social cognitive deficits of schizophrenia,
2. test the efficacy of OT in normalizing the neural abnormalities underlying these social deficits, and
3. develop and optimize novel treatments for these currently untreatable deficits.

ELIGIBILITY:
Inclusion Criteria for Patients:

* 18-40 years of age
* Male
* Must comprehend English
* Meet DSM-IV criteria for schizophrenia, schizophreniform or schizoaffective disorder
* None or only minor changes to medications in the past week
* Able to use nasal spray
* Must be capable of providing informed consent
* Clinically stable

Inclusion Criteria for Healthy Controls:

* 18-40 years of age
* Male
* Must comprehend English
* No diagnosis of mental disorder according to DSM-IV TR
* Able to use nasal spray
* Must be capable of providing informed consent
* Clinically stable

Exclusion Criteria:

* Female
* Active substance abuse or dependence as determined by a Urine Toxicology Drug Screening
* DSM-IV diagnosis of any disorder other than schizophrenia
* Medical conditions (atrophic rhinitis, recurrent nose bleeds and cranial surgical procedures (hypophysectomy), congestion or sinus problems that could interfere with the study as per the opinion of the investigator
* Hearing deficits
* A pacemaker, extensive dental work, or any magnetic metal implants
* Any history of severe brain trauma

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in MEG neural activation patterns | Oxytocin and placebo administration days at least 1-week apart
  During tasks in which participants will see and hear various stimuli, investigators will measure the change in neural activity in the amygdala, the dorsal anterior cingulate cortex, as well as the fusiform gyrus using the MEG scanner.

SECONDARY OUTCOMES:
Change in performance on Facial Recognition Task | Oxytocin and placebo administration days at least 1-week apart
  In the Facial Recognition Task, subjects will be presented with various computerized emotional stimuli and will be asked to make a choice. Participants will then respond to the stimuli by pressing a either left or right on the control box and their reaction time will be measured.
Change in performance on International Affective Picture System (IAPS) task | Oxytocin and placebo administration days at least 1-week apart
  In the IAPS Tasks, subjects will view images of people, objects, and scenes from the IAPS (International Affective Picture System). Participants will then respond by pressing a either left or right on the control box to chose a number from 1 (i.e. least disturbing) to 9 (i.e. most disturbing) and their reaction time will be measured.
UCLA Loneliness Scale | 1 day
  The UCLA Loneliness Scale assesses the loneliness level of participants. It is a 20-item scale where responses are measured from O ("I often feel this way") to N ("I never feel this way").
Experiences in Close Relationships-Relationship Structures (ECR-RS) Questionnaire | 1 day
  The ECR is used to evaluate the construct of adult attachment. The scale involves 36 itemized statements split into four parts, each part referring to a different attachment figure. Participants rank each item using a 7-point likert scale.
Childhood Trauma Questionnaire (CTQ) | 1 day
  The CTQ is a brief survey of 6 early traumatic experiences, including death, divorce, violence, sexual abuse, illness or other. The scale determines and assesses an individual's understanding of their childhood trauma, if applicable.
Parental Bonding Instrument (PBI) | 1 day
  The PBI measures fundamental parenting styles as perceived the child. The questionnaire is retrospective in that it asks the adult participant to answer the questions based on how they remember their parents to be during up until they were 16 years old. The measure is completed for both mothers and fathers separately. There are 25 questions where half the questions are focused on how the parent cared for them and half are focused on how the parents protected them. A likert scale is used to measure responses where 1 is agree (i.e. very like) and 4 is disagree (i.e. very dislike).
Emotional Quotient Scale (EQS) | 1 day
  The EQ is a 60-item self-report questionnaire that is designed to measure empathy in adults. Participants use a 4 item likert scale to record their responses (1=definitely agree, 4= definitely disagree).
Fagerstom Nicotine Dependence Test | 1 day
  The FNDT is the standard measure of an individual's physical addiction to nicotine. The test contains six items to evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.
Quality of Life Scale (QLS) | 1 day
  The QLS is a 21-item clinical rating scale where the interviewer rates the participant's responses on a scale of 1-6 where 6 indicates no impairment. In this study, an abbreviated version of the QLS is used that includes 9 of the 21 items. The 9 items are each derived from the sections examining interpersonal relations, occupational role functioning, intrapsychic foundations, and common objects.
Social Functioning Scale (SFS) | 1 day
  The SFS is designed to assess a subject's social skills and performance, and to measure functions that are of importance for schizophrenic patients. It is a 79-item scale completed by the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Josh D Woolley, MD/PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (1):
- University of California, San Francisco, San Francisco, California, United States